CLINICAL TRIAL: NCT00125619
Title: Internally v. Externally Guided BWSTT for Locomotor Recovery Post-stroke
Brief Title: Internally Versus Externally Guided Body Weight-Supported Treadmill Training (BWSTT) for Locomotor Recovery Post-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B4032-I
Record Dates: First submitted 2005-07-28; First posted 2005-08-01 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2016-12

CONDITIONS: Stroke
Keywords: biomechanics; stroke; electromyography; Gait disability stroke; locomotor therapy; muscular weakness; reflex variability stroke
MeSH Terms: conditions — Stroke; Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Therapist assisted (Active Comparator): Therapist assisted locomotor training (partial body-weight supported)
  Interventions: Behavioral: Locomotor training
- Arm 2: Robot-assisted (Experimental): Robot-assisted locomotor training (partial body-weight supported)
  Interventions: Behavioral: Locomotor training

INTERVENTIONS:
Behavioral: Locomotor training — This study compares two forms of Iocomotor training: 1) standard or manual - in which an individual is provided partial body weight support while walking on a treadmill with assistance of 1-3 therapists to move the legs and stabilize the trunk/pelvis and 2) robotic-guided - in which an exoskeleton robot (Lokomat) guides movement of the walking pattern. Partial body-weight support, treadmill walking and treadmill speed are consistent between the study arms.
  Other Names: partial body-weight supported treadmill training, body-weight supported treadmill training

SUMMARY:
The overriding goal of this proposal is to identify the critical physiological and biomechanical effects of BWSTT for promoting improved locomotor function in persons with post-stroke hemiparesis.

DETAILED DESCRIPTION:
In this pilot study, we tested two forms of locomotor training for gait rehabilitation in persons post-stroke: traditional locomotor training (partial body-weight support and manual assistance of therapists) vs. robotic-assisted locomotor training (partial body-weight support and robotic guidance with the Lokomat). We enrolled 16 persons with chronic (>6 months) hemiparesis post-stroke who were randomized to traditional/manual or robotic locomotor training. All individuals received 12 sessions (thrice weekly for four weeks) of training. Each session involved 30 minutes of stepping.

The complete study results are published.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cerebrovascular accident
* Single event
* Unilateral hemiplegia
* Locomotor disability
* Ability to walk independently 25' on level ground (may use an assistive device [cane or walker]; may NOT use a brace)
* Cognitive ability to follow 3-step commands

Exclusion Criteria:

* Unstable or uncontrolled blood pressure
* Uncontrolled seizures
* Severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolynn Patten, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States

REFERENCES:
- [Result] Westlake KP, Patten C. Pilot study of Lokomat versus manual-assisted treadmill training for locomotor recovery post-stroke. J Neuroeng Rehabil. 2009 Jun 12;6:18. doi: 10.1186/1743-0003-6-18. PMID 19523207
- [Result] Spiess MR, Jaramillo JP, Behrman AL, Teraoka JK, Patten C. Unexpected recovery after robotic locomotor training at physiologic stepping speed: a single-case design. Arch Phys Med Rehabil. 2012 Aug;93(8):1476-84. doi: 10.1016/j.apmr.2012.02.030. Epub 2012 Mar 23. PMID 22446153

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 2: Robot-assisted: Rehabilitation got Post-stroke Hemiparesis
  Robotic-driven Locomotor Training for Gait (a robotic device called the Lokomat guides the participant's legs during locomotion over a treadmill with partial body weight support).
- Arm 1: Therapist Assisted: Rehabilitation for Post-Stroke hemiparesis Body-weight Supported Locomotor Training (manual, with therapist assistance for movement of the paretic leg)
Period: Overall Study
Arm/Group | Arm 2: Robot-assisted | Arm 1: Therapist Assisted
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 2: Robot-assisted: Rehabilitation for Post-stroke Hemiparesis
  Robotic-driven Locomotor Training for Gait (a robotic device called the Lokomat guides the participant's legs during locomotion over a treadmill with partial body weight support).
- Total: Total of all reporting groups
Arm/Group | Arm 2: Robot-assisted | Arm 1: Therapist Assisted | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (16.9) | 55.1 (13.6) | 56.8 (14.4)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
Self-selected Overground Walking speed [Mean (Standard Deviation); unit: meters per second] | 0.62 (0.31) | 0.62 (0.28) | 0.62 (0.28)
Fast Walking Speed [Mean (Standard Deviation); unit: meters per second] | 0.87 (0.55) | 0.72 (0.37) | 0.80 (0.47)
Six Minute Walk Test [Mean (Standard Deviation); unit: distance walked, meters] | 267.3 (187.2) | 234.3 (141.2) | 250.8 (161.1)
Step-length Asymmetry [Mean (Standard Deviation); unit: ratio] — Measure is a ratio of paretic/non-paretic step length calculated as follows:
  = ABS[1-(paretic step length/non-paretic step length)]
  Values approaching 0 reveal greater symmetry.
  ratio | 0.53 (0.58) | 0.39 (0.37) | 0.45 (0.48)
Lower Extremity Fugl-Meyer Motor Assessment [Mean (Standard Deviation); unit: units on a scale] — The Fugl-Meyer Motor Assessment is a standardized clinical assessment used to determine the magnitude of motor impairment (or severity) following stroke. There are separate scales for the upper and lower extremities. Here we used the lower extremity component which has a range of 36 points. Higher scores reflect better motor status than lower scores. Importantly, there is a remarkable ceiling effect with the FMA, thus a full score of 36 points does not indicate an individual post-stroke has fully recovered.
  units on a scale | 23.0 (4.3) | 21.4 (5.1) | 23 (4.5)
Short Physical Performance Battery [Mean (Standard Deviation); unit: units on a scale] — The Short Physical Performance Battery measures 3 components of physical function: walking speed, strength - assessed through repeated sit-to-stand movements, and balance. The SPPB is scored over a range of 0-12 points, where 12 is the highest, or best, score. Each of the 3 components contributes 4 points to the total SPPB, although sub-scores are not typically calculated and/or interpreted.
  units on a scale | 6.9 (3.4) | 7.8 (3.0) | 7.31 (3.1)
Berg Balance Scale [Mean (Standard Deviation); unit: units on a scale] — The Berg Balance Scale is a standardized clinical assessment of balance function involving performance of 14 tasks ranging from sitting unsupported to standing on one leg with eyes closed. It is scored on a range of 0 - 56 points where 56 is the best score, which is generally equivalent to normal.
  units on a scale | 46.9 (7.5) | 47 (7.0) | 46.9 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Self-selected Overground Walking Speed
Description: Overground walking speed determined as rate of walking over a 10 meter distance.
Time Frame: 4 weeks (s/p 12 sessions of locomotor training)
Measure: Mean (Standard Deviation); unit: meters/s
Arm/Group | Arm 2: Robot-assisted | Arm 1: Therapist Assisted
Number analyzed (Participants) | 8 | 8
meters/s | 0.72 (0.38) | 0.65 (0.29)
Statistical Analysis 1: Comparison: Arm 2: Robot-assisted vs Arm 1: Therapist Assisted; Between group comparison of Robot (Lokomat) vs. Manual (therapist-assisted) training; Test type: Superiority or Other; p = 0.72, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm 2: Robot-assisted; Within group test for change pre- vs. post-training due to Robot (Lokomat) training; Test type: Superiority or Other; p < .05, Wilcoxon Signed Ranks
Statistical Analysis 3: Comparison: Arm 1: Therapist Assisted; Within group test for change pre- vs. post-training due to Manual (Therapist Assisted) training; Test type: Superiority or Other; p > .05, Wilcoxon Signed Ranks

2. Secondary Outcome: Fast Walking Speed
Description: Fastest comfortable walking speed measured while walking overground
Time Frame: 4 weeks (s/p 12 training sessions)
Measure: Mean (Standard Deviation); unit: meters/s
Arm/Group | Arm 2: Robot-assisted | Arm 1: Therapist Assisted
Number analyzed (Participants) | 8 | 8
meters/s | 0.96 (0.66) | 0.70 (0.33)
Statistical Analysis 1: Comparison: Arm 2: Robot-assisted vs Arm 1: Therapist Assisted; Between-groups comparison of Robot vs. Manual training; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm 1: Therapist Assisted; Within groups comparison (pre- vs. post-treatment) due to Manual (therapist-assisted) treatment; Test type: Superiority or Other; p > .05, Wilcoxon Signed Ranks
Statistical Analysis 3: Comparison: Arm 2: Robot-assisted; Within-groups comparison of pre- vs. post-treatment effects for Robot (Lokomat) training; Test type: Superiority or Other; p < .05, Wilcoxon Signed Ranks

3. Secondary Outcome: Six Minute Walk
Description: distance, in meters, walked overground over a six minute interval.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Arm 2: Robot-assisted | Arm 1: Therapist Assisted
Number analyzed (Participants) | 8 | 8
meters | 278.1 (176.5) | 212.4 (113.5)
Statistical Analysis 1: Comparison: Arm 2: Robot-assisted vs Arm 1: Therapist Assisted; Between-groups comparison of robot vs. manual training; Test type: Superiority or Other; p > .05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm 1: Therapist Assisted; Within group comparison of pre- vs. post-treatment effects for manual training; Test type: Superiority or Other; p > .05, Wilcoxon Signed Ranks
Statistical Analysis 3: Comparison: Arm 2: Robot-assisted; Within group comparison of pre- vs. post-treatment effects of robot training; Test type: Superiority or Other; p > .05, Wilcoxon signed ranks

4. Secondary Outcome: Step Length Ratio (Abs)
Description: measure of step length symmetry, calculated as = ABS [1 - (Pstep length / NPstep length)]
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Arm 2: Robot-assisted | Arm 1: Therapist Assisted
Number analyzed (Participants) | 8 | 8
ratio | 0.37 (0.46) | 0.34 (0.35)
Statistical Analysis 1: Comparison: Arm 2: Robot-assisted vs Arm 1: Therapist Assisted; Between groups comparison of effects of robot vs. manual training; Test type: Superiority or Other; p > .05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm 1: Therapist Assisted; Within groups comparison of pre- vs. post-treatment effects of manual training; Test type: Superiority or Other; p > .05, Wilcoxon Signed Ranks
Statistical Analysis 3: Comparison: Arm 2: Robot-assisted; Within group comparison of pre- vs. post-training effects of robot training; Test type: Superiority or Other; p < .05, Wilcoxon Signed Ranks

5. Secondary Outcome: Lower Extremity Fugl-Meyer Motor Assessment
Description: Standardized clinical measure of motor impairment. The lower extremity (leg) sub-scale ranges from 0 - 35 points, where less impairment corresponds with scores approaching 35 and worse impairment corresponds with scores approaching 0.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2: Robot-assisted | Arm 1: Therapist Assisted
Number analyzed (Participants) | 8 | 8
units on a scale | 25.6 (5) | 22.4 (5.2)
Statistical Analysis 1: Comparison: Arm 2: Robot-assisted vs Arm 1: Therapist Assisted; Between groups comparison of robot vs. manual training; Test type: Superiority or Other; p > .05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm 1: Therapist Assisted; Within groups comparison for pre- vs. post-training effects of manual training; Test type: Superiority or Other; p > .05, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Arm 2: Robot-assisted; Within group comparison for pre- vs. post-training effects of robot training; Test type: Superiority or Other; p > .05, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Short Physical Performance Battery
Description: Standardized clinical measure of physical function involving tests of: walking speed, strength (repeated chair rise), and balance. The scale ranges from 0 - 12 points with better physical function as the score approaches 12 points and worse physical function as the score approaches 0 points.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2: Robot-assisted | Arm 1: Therapist Assisted
Number analyzed (Participants) | 8 | 8
units on a scale | 7.9 (3.2) | 8.5 (3.1)
Statistical Analysis 1: Comparison: Arm 2: Robot-assisted vs Arm 1: Therapist Assisted; Between groups comparison of robot vs. manual training; Test type: Superiority or Other; p > .05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm 1: Therapist Assisted; Within group comparison of pre- vs. post-training effects of manual training; Test type: Superiority or Other; p > .05, Wilcoxon Signed Ranks
Statistical Analysis 3: Comparison: Arm 2: Robot-assisted; Within group comparison of pre- vs. post-treatment effects of robot training; Test type: Superiority or Other; p < .05, Wilcoxon Signed Ranks

7. Secondary Outcome: Berg Balance Scale
Description: Clinical measure of balance
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2: Robot-assisted | Arm 1: Therapist Assisted
Number analyzed (Participants) | 8 | 8
units on a scale | 48.3 (6.8) | 51.0 (5.4)
Statistical Analysis 1: Comparison: Arm 2: Robot-assisted vs Arm 1: Therapist Assisted; Between groups comparison of robot vs. manual training; Test type: Superiority or Other; p > .05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm 1: Therapist Assisted; Within group comparison of pre- vs. post-training effects of manual training; Test type: Superiority or Other; p < .05, Wilcoxon Signed Ranks
Statistical Analysis 3: Comparison: Arm 2: Robot-assisted; Within group comparison of pre- vs. post-treatment effects of robot training; Test type: Superiority or Other; p < .05, Wilcoxon Signed Ranks

ADVERSE EVENTS:
Groups:
- ARM2: Rehabilitation got Post-stroke Hemiparesis
  Robotic-driven Locomotor Training for Gait (a robotic device called the Lokomat guides the participant's legs during locomotion over a treadmill with partial body weight support).
- Arm 1: Rehabilitation for Post-Stroke hemiparesis Body-weight Supported Locomotor Training (manual, with therapist assistance for movement of the paretic leg)
Arm/Group | ARM2 | Arm 1
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Small sample size, but consistent with intent of pilot study Inclusion criterion was >6 months post-event, allowing for large heterogeneity in chronicity Intervention was limited (12 sessions distributed over 4 weeks)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No